CLINICAL TRIAL: NCT06240312
Title: Optic Nerve Head Strain as Biomarker for Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00431247
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All subjects (Other): Each subject will be imaged at two different times and eye pressures
  Interventions: Device: Images of eye at 2 eye pressures

INTERVENTIONS:
Device: Images of eye at 2 eye pressures — subject images of the eye's optic nerve head are studied

SUMMARY:
The investigators will test the hypothesis that images of the optic nerve head taken a 2 different eye pressures will yield strain estimates that are predictive of the course of glaucoma.

DETAILED DESCRIPTION:
Existing glaucoma patients and suitable control adults will be imaged with an FDA-approved optical coherence tomography instrument. Those who are imaged at 2 different eye pressures will generate biomechanical strain estimates. These will be compared to visual field and retinal nerve fiber layer measurements over time. The investigators expect that baseline strain and their changes over time will be associated with progression rate of glaucoma damage, providing a biomarker for susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Existing glaucoma patients of Johns Hopkins

Exclusion Criteria:

* Inability to perform imaging
* illiterate
* hearing impaired
* non-English speakers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Optic nerve head mechanical strain compared to visual field change over time | Approximately 3 years
  Strains measured at baseline are tested for association with glaucoma course

CONTACTS AND LOCATIONS:
Overall Officials: Harry Quigley, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No